CLINICAL TRIAL: NCT04781712
Title: Feasibility of a Modular mHealth for Tailored Rehabilitation During the Treatment of Breast Cancer
Brief Title: Feasibility of a Modular mHealth for Tailored Rehabilitation of Breast Cancer
Acronym: MMHTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMC-2018-10-062
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management using mHealth (Experimental): Self-management (physical activity, sleep, exercise, education, etc.) using mHealth
  Interventions: Behavioral: Modular mHealth for Tailored Rehabilitation
- Exercise using brochure (No Intervention): Only exercise using brochure

INTERVENTIONS:
Behavioral: Modular mHealth for Tailored Rehabilitation — an individually tailored self-management through the mHealth app with a smart band worn on the wrist
  Other Names: mHealth
  Arms: Self-management using mHealth

SUMMARY:
This study investigated the feasibility of the novel modular mobile health (mHealth) for personalized rehabilitation and explored the participants' satisfaction and app data during treatment of breast cancer.

DETAILED DESCRIPTION:
This is prospective, feasible, parallel study in post-operative patients with breast cancer and during treatment. Disability of Arm, Shoulder, Hands (DASH), Physical activity data (IPAQ-SF), Physical measurement such as hand grip strength, body mass index (BMI), muscle mass, and differences in arm circumference, PRO-CTCAE, Distress Thermometer, needs and satisfaction in app, personal health record of app (exercise, daily step count, etc.) Measure will be evaluated on 1-month, 2-month, 4-month, 6-month, 9-month, and 12-month after POD.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer at TNM stage 0 ~ III
* Patients who will undergo the treatment (chemotherapy, radiation therapy, and hormone therapy) after surgery
* Patients who had a mobile phone (Android or iOS)

Exclusion Criteria:

- Patients who have metastases or recurrence to other organs were excluded

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
satisfaction score in app contents | 1 to 12month
  satisfaction score in app contents, Likert scale (5-point, higher scores mean a better)
Needs score in app contents | 1 to 12month
  Needs score in app contents, Likert scale (5-point, higher scores mean a better)
DASH (Disabilities of Arm, Shoulder, Hands) | 1 month, 2month, 4month, 6month, 9month, 12month
  Change from Baseline DASH score at 12 months, higher scores mean a worse (0-100)

SECONDARY OUTCOMES:
Physical measurement (handgrip strength) | 1 to 12month
  Handgrip strength (kg)
Physical measurement (of body composition, BMI) | 1 to 12month
  Body mass index
Physical measurement (of body composition, muscle mass) | 1 to 12month
  muscle mass
Physical measurement (upper extremity volume) | 1 to 12month
  differences in arm circumference
Physical activity (IPAQ-SF Questionnaire) | 1 to 12month
  Total METs within recent 7 days (vigorous, moderate, walking, sitting), higher values mean a better
PRO-CTCAE (patients reported outcomes) | 1 to 12month
  Symptoms during treatment
Distress thermometer (distress level) | 1 to 12month
  Distress level during treatment, higher scores mean a worse (0-10)
App use data (personal health record)_Exercise compliance rate | 1 to 12month
  Exercise time, higher values mean a better
App use data (personal health record)_Physical activity change | 1 to 12month
  daily step count (number), higher values mean a better physical activity
App use data (personal health record)_interest of contents | 1 to 12month
  contents view (number), higher values mean a better compliance rate
App use data (personal health record)_sleep | 1 to 12month
  sleep compliance rate (%), higher values mean a better compliance rate

CONTACTS AND LOCATIONS:
Overall Officials: JIHYE HWANG, Professor, Study Chair — Physical & Rehabilitation Medicine Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided